CLINICAL TRIAL: NCT04944641
Title: Epilepsy Prevalence and Intervention Study in Zhejiang Province, China
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Hangzhou Center of Disease Control and Prevention (Other Government); The Central Hospital of Lishui City (Other); The Second Affiliated Hospital of Jiaxing University (Other); Zhejiang University (Other); Children's Hospital Affiliated to Zhejiang University School of Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2013-032
Record Dates: First submitted 2021-06-08; First posted 2021-06-29 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Epilepsy
Keywords: epilepsy prevalence, intervention
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Intervention Model Description: randomly group into two

ARMS (2):
- A: Routine AED group (Experimental): Routine and proper antiepileptic drugs group
  Interventions: Drug: routine and proper antiepileptic drugs
- B: AED and education group (Experimental): Routine, proper antiepileptic drugs and education group
  Interventions: Behavioral: education on epilepsy; Drug: routine and proper antiepileptic drugs

INTERVENTIONS:
Behavioral: education on epilepsy — education on epilepsy, including epilepsy diary, pamphlet，discussion between patients and phone visits and so on
  Arms: B: AED and education group
Drug: routine and proper antiepileptic drugs — routine and proper antiepileptic drugs

SUMMARY:
To carry out the epidemiological investigation on epilepsy in Zhejiang Province, China, and then establish early comprehensive intervention to help patients with epilepsy to improve seizure control and the quality of life.

DETAILED DESCRIPTION:
To carry out the epidemiological investigation on epilepsy in Zhejiang Province, China, and then establish early comprehensive intervention（proper antiepileptic drugs and education intervention） to help patients with epilepsy to improve seizure control and the quality of life.

ELIGIBILITY:
Inclusion Criteria:

Newly diagnosed and untreated epilepsy; Aged 14 and above; Sign the informed consents.

Exclusion Criteria:

With intellectual development disorder; With serious heart and lung diseases.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-09-13 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline seizures frequency 1 | 12 months
  change from baseline seizures frequency at 12 months, seizure frequency is defined as the number of seizure attacks during 3 months before baseline or endpoint)
Change from baseline seizures frequency 2 | 24 months
  change from baseline seizures frequency at 24 months, seizure frequency is defined as the number of seizure attacks during 3 months before baseline or endpoint)
Occurrence of refractory epilepsy | 24 months
  occurrence of refractory epilepsy at 24 months

SECONDARY OUTCOMES:
Quality of life (QOL scales) | 2 year
  Quality of Life Scale, high scores mean a better outcome

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang
  - Shengzhou People's Hospital, Shengzhou